CLINICAL TRIAL: NCT04823897
Title: A Phase 1 Open-Labelled, Single-Arm, Dose-Escalation, Clinical and Pharmacology Study of CCI-001 in Patients With Recurrent and/or Metastatic Solid Tumours
Brief Title: A Study of CCI-001 in Patients With Recurrent and/or Metastatic Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMatrix Holdings Ltd (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PMH-001
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cancer: Recurrent and/or Metastatic Solid Tumours

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm, single-center, Phase I dose-escalation study of CCI-001 in patients with recurrent and/or metastatic solid tumours.
  Patients will be treated in cohorts of 3, with the starting cohort having an assigned dose of CCI-001 of 1.2 mg/m2. If safety criteria are met, subsequent cohorts will be administered escalating doses of CCI-001, using the modified accelerated dose-escalation method.
  Any cohort in which a patient experiences DLT in Cycle 1 will be expanded to 6 patients. Dose escalation will continue if only 1 of 6 patients in a cohort experiences DLT. If 2 patients within a cohort experience DLT, the maximum tolerated dose will have been reached/exceeded.
  The cohort at the dose below this cohort will be expanded to 6 patients to ensure tolerability. If none of the 3 additional patients at this lower dose experiences DLT, that dose will be declared as the recommended dose for the dose expansion phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): Dose escalation phase: CCI-001 will be administered at the starting dose to a cohort of patients with recurrent and/or metastatic solid tumours. The dose will be escalated sequentially in subsequent cohorts to determine the maximum tolerated dose, or recommended dose for the dose expansion cohort.
  Dose expansion phase: patients with the following tumour types will be permitted to enroll: transitional cell bladder cancer, pancreaticobiliary adenocarcinomas, gynecologic cancers (ovarian, cervical, endometrial), and lung adenocarcinoma. These patients will be treated at the dose determined during the dose escalation phase.
  Interventions: Drug: CCI-001

INTERVENTIONS:
Drug: CCI-001 — Dose Escalation Phase: CCI-001 will be administered by intravenous infusion starting at 1.2mg per square metre of body surface area in the first cohort. The dose will be escalated sequentially in subsequent cohorts. The degree of dose escalation between subsequent cohorts will depend on tolerability, as judged by NCI-CTCAE grading. Once the maximum tolerated dose is determined this phase will be complete.
  Dose Expansion Phase: cohorts of patients with the following tumour types will be enrolled: transitional cell bladder cancer, pancreaticobiliary adenocarcinomas, gynecologic cancers (ovarian, cervical, endometrial), and lung adenocarcinoma. These patients will be treated at the dose determined in the dose escalation phase.

SUMMARY:
CCI-001 is a novel colchicine derivative that is being developed by PharmaMatrix Holdings Ltd. (PharmaMatrix). The drug binds to tubulin, a component of the microtubule polymers which are required for a wide range of cellular processes, perhaps most importantly, cell division and mitosis. CCI-001 has been shown to bind more strongly to β-III tubulin, a tubulin subtype which is overexpressed in many cancers.

This trial is being undertaken as a first-in-human, Phase I trial in patients with recurrent and/or metastatic solid tumours. Primary Objectives are to examine the compound's safety profile, and to determine the recommended dose. Secondary Objectives are to determine the compound's pharmacokinetic parameters and to evaluate the clinical response rate and survival. Expansion cohorts in in tumour types known to be sensitive to other approved agents with similar mechanism of action will be treated at the recommended dose: transitional cell bladder cancer, pancreaticobiliary adenocarcinomas, gynecologic cancers (ovarian, cervical, endometrial), and lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent/assent prior to initiation of any study-specific activities/procedures.
2. Dose escalation phase: Patients must have histologically or cytologically confirmed recurrent or metastatic solid tumours. Patients must have disease progression on the last treatment exposed to, have exhausted available approved lines of therapy or better-characterized therapies that, at the discretion of the investigator, is felt to be more appropriate therapy, or have malignancies for which there are no approved therapies.

   Dose expansion phase: patients with the following tumour types will be permitted to enroll: transitional cell bladder cancer, pancreaticobiliary adenocarcinomas, gynecologic cancers (ovarian, cervical, endometrial), and lung adenocarcinoma.
3. Four weeks must have elapsed since prior chemotherapy, hormonal therapy, targeted therapy, or radiation therapy. There is no restriction in the amount of bone marrow previously radiated.
4. Recovery to baseline or grade 1 for all drug-related toxicities due to prior chemotherapy, radiation, hormonal therapy, or molecular targeted therapy, except for alopecia.
5. Age ≥18 years.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤1.
7. Life expectancy of greater than 12 weeks.
8. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count ≥ 1.5 x 10^9/L
   * hemoglobin ≥ 90 g/L
   * platelets ≥ 100 x 10^9/L
   * total bilirubin ≤ 1.5 X upper limit of normal (ULN)
   * AST(SGOT) and ALT(SGPT) ≤ 2.5 X ULN (≤ 5 X ULN in the presence of liver metastases)
   * Creatinine (Cr) ≤ 1.5 X ULN
9. Cardiac ejection fraction by echocardiogram must be >50% at baseline. Any structural changes found must be reviewed by the treating investigator and deemed acceptable and safe prior to study enrolment. Any noted cardiac fibrosis will exclude a patient.
10. Baseline ECG with QTc ≤ 470msec for females and ≤ 450msec for males.
11. Agree to use adequate contraception for the duration of study participation and for 12 months after receiving the final dose of study drug.
12. Ability and willingness to adhere to study required procedures.
13. Patient must have measurable disease according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria.

Exclusion Criteria:

1. Patients may not be receiving any other investigational agents, chemotherapy, immunotherapy, radiotherapy, or molecular targeted agents within 28 days prior to enrollment to study unless discussed with the Principal Investigator.
2. Patients may not have symptomatic central nervous system (CNS) metastases. Patients with treated CNS metastases are eligible, provided their disease is radiographically stable over a period of ≥ 8 weeks, asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants for the treatment of the symptoms from their brain metastases. Screening of asymptomatic patients without a history of CNS metastases is not required.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to CCI-001 such as derivatives of colchicine.
4. The presence of grade 2 or higher peripheral neuropathy due to prior medical condition (such as multiple sclerosis), medications, or other etiologies.
5. Any psychological, familial, sociological, or geographical conditions that do not permit medical follow-up and compliance with the study protocol.
6. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant or nursing women.
8. Human Immunodeficiency Virus (HIV)-positive patients.
9. Hepatitis B- and/or C-positive patients. A negative test is required at screening.
10. History of other invasive cancer within 2 years of study entry. The exceptions are in situ cervical cancer, basal cell carcinoma or squamous cell carcinoma of the skin, and localized prostate cancer after curative therapy such as surgery, or radiation (Gleason score ≤ 7). For these exceptions, all treatment must have been completed 6 months prior to enrollment.
11. Patients taking warfarin. Low-dose or therapeutic dose of heparin or low-molecular weight heparin are allowed.
12. Cardiac fibrosis on echocardiogram. Adherence to all inclusion and exclusion criteria is mandatory; no waivers will be granted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of intravenously infused CCI-001 in patients with recurrent and/or metastatic solid tumours by determining the dose-limiting toxicity (DLT) of the compound. | Cycle 1 (28 days)
  DLT in this study will be determined against a pre-defined set of criteria based on the NCI-CTCAE v. 5.0 grading system.
To determine, during the dose escalation phase, the recommended dose of intravenously infused CCI-001 for the dose expansion phase of the trial. | Cycle 1 (28 days)
  The recommended dose will be the dose level below that for the cohort in which maximum tolerated dose (MTD) was reached/exceeded. MTD will have been reached when 2 or more patients in a cohort experience DLT.

SECONDARY OUTCOMES:
To evaluate the clinical response rate in patients treated with CCI-001 with recurrent and/or metastatic solid tumours, with particular attention to those in expansion cohorts | Patients will have a baseline scan prior to dosing, and re-evaluated with imaging every 8 weeks. To continue from baseline scan to first documented date of disease progression, or date of death from any cause, to a maximum of 36 months.
  All patients with measurable disease will be assessed by standard criteria. Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria will be utilized to determine response based on CT and/or MRI scans.
To evaluate survival in patients treated with CCI-001 with recurrent and/or metastatic solid tumours, with particular attention to those in expansion cohorts | Start of treatment period (Cycle 1, Day1) to 30 days past the last treatment. Each Cycle is 28 days.
  Descriptive statistics will be utilized to evaluate patient survival.
To determine the time to maximum plasma level (Tmax) of CCI-001 administered intravenously. | Measured on Cycle 1 Days 1 and 15, Cycle 2 Day 1 (Each cycle is 28 days)
  Tmax is the time at which the maximum plasma CCI-001 concentration is achieved.
To determine the maximum plasma concentration (Cmax) of CCI-001 administered intravenously. | Measured on Cycle 1 Days 1 and 15, Cycle 2 Day 1 (Each cycle is 28 days)
  Cmax is the maximum plasma CCI-001 concentration that is achieved post administration.
To determine the area under the curve (AUC) of CCI-001 administered intravenously. | Measured on Cycle 1 Days 1 and 15, Cycle 2 Day 1 (Each cycle is 28 days)
  AUC is the measure of total CCI-001 exposure after administration.
To determine the terminal half life (t1/2) of CCI-001 administered intravenously. | Measured on Cycle 1 Days 1 and 15, Cycle 2 Day 1 (Each cycle is 28 days)
  t1/2 is the measure of the time it takes CCI-001 plasma concentration to decrease by 50%, after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Spratlin, MD, Principal Investigator — Alberta Health Services, University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No